CLINICAL TRIAL: NCT03783130
Title: VRC 018: A Phase I Dose Escalation, Randomized, Open-Label Clinical Trial to Evaluate Dose, Safety, Tolerability and Immunogenicity of a HIV-1 Vaccine, VRC-HIVRGP096-00-VP, With Alum in Healthy Adults
Brief Title: Dose, Safety, Tolerability, and Immunogenicity of an HIV-1 Vaccine, VRC-HIVRGP096-00-VP, With Alum in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 190031; 19-I-0031
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Human Immunodeficiency Virus Prevention; Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus; Immune Response; Neutralizing Antibodies; HIV Prevention; Cellular Immunogenicity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Aluminum Hydroxide; aluminum sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Trimer 4571 (100 mcg) IM with alum (Experimental): Trimer 4571 injections (100 mcg), with 500 mcg of alum field mixed, administered intramuscularly (IM) in a 1 mL volume by Needle/Syringe on Day 0, Week 8, and Week 20
  Interventions: Biological: VRC-HIVRGP096-00-VP; Other: Alum Adjuvant
- Group 2: Trimer 4571 (100 mcg) SC with alum (Experimental): Trimer 4571 injections (100 mcg), with 500 mcg of alum field mixed, administered subcutaneously (SC) in a 1 mL volume by Needle/Syringe on Day 0, Week 8, and Week 20
  Interventions: Biological: VRC-HIVRGP096-00-VP; Other: Alum Adjuvant
- Group 3: Trimer 4571 (500 mcg) IM with alum (Experimental): Trimer 4571 injections (500 mcg), with 500 mcg of alum field mixed, administered intramuscularly (IM) in a 1 mL volume by Needle/Syringe on Day 0, Week 8, and Week 20
  Interventions: Biological: VRC-HIVRGP096-00-VP; Other: Alum Adjuvant
- Group 4: Trimer 4571 (500 mcg) SC with alum (Experimental): Trimer 4571 injections (500 mcg), with 500 mcg of alum field mixed, administered subcutaneously (SC) in a 1 mL volume by Needle/Syringe on Day 0, Week 8, and Week 20
  Interventions: Biological: VRC-HIVRGP096-00-VP; Other: Alum Adjuvant

INTERVENTIONS:
Biological: VRC-HIVRGP096-00-VP — Trimer 4571 drug product is an investigational HIV vaccine which mimics the native HIV-1 envelope complex. This soluble HIV-1 envelope product consists of an HIV-1 envelope (Env) trimer variant, derived from clade A, strain BG505, with stabilizing mutations and engineered disulfide bonds, specifically recognized by broadly neutralizing antibodies and resists gp120 conformational change caused by CD4 binding.
  Other Names: Trimer 4571
Other: Alum Adjuvant — Adjuvant is an aluminum hydroxide suspension (alum) mixed with Trimer 4571 to improve the immune response to the investigational vaccine.
  Other Names: Aluminum Hydroxide Suspension; Alum

SUMMARY:
Background:

HIV stands for human immunodeficiency virus, which is the virus that causes AIDS. There is currently no licensed vaccine to prevent HIV infection. Researchers want to test a vaccine called Trimer 4571 for the first time. It was made at the National Institutes of Health (NIH) and contains no HIV. The vaccine is mixed with a substance called alum and injected in the arm. Alum is included to boost the body's immune response to the vaccine. It has been used in licensed vaccines for over 60 years and has been found to be safe.

Objectives:

To see if the vaccine Trimer 4571 is safe, well-tolerated, and to study immune responses to it.

Eligibility:

Healthy adults ages 18-50 years

Design:

Participants were screened with a physical exam and blood tests. They agreed to not become pregnant and to avoid behavior that would put them at high-risk for HIV infection during the study.

Participants had about 15 study visits over about 9 months.

The first 6 participants received a low dose of the vaccine mixed with alum.

Once the low dose was deemed safe, 10 new participants were allocated to receive a higher dose.

All participants were randomly assigned to get the vaccine by injection in a muscle or under the skin.

All participants received a total of 3 vaccine injections over 20 weeks. Each visit where participants received the vaccine lasted about 5 hours. Participants were watched after each injection. Participants who were able to get pregnant would have a pregnancy test before each injection.

Participants received a thermometer and recorded their temperature and symptoms every day for 1 week after each injection. The injection site was checked for redness, swelling, or bruising.

At follow-up visits, participants had blood drawn and checked for health changes or problems. Follow up visits lasted about 1-2 hours.

DETAILED DESCRIPTION:
Design:

This is a Phase I, open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of VRC-HIVRGP096-00-VP (Trimer 4571) with aluminum hydroxide suspension (alum) as adjuvant in a three-injection regimen. The hypotheses were that the vaccine will be safe and tolerable and will induce detectable immune responses. The primary objective was to evaluate the safety and tolerability of the investigational vaccine at three doses administered with alum. Secondary objectives were to evaluate humoral and cellular immunogenicity of the investigational vaccine regimens.

Study Product:

VRC-HIVRGP096-00-VP (Trimer 4571) was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID). The soluble HIV-1 envelope product consists of an HIV-1 envelope (Env) trimer variant, derived from clade A, strain BG505, with stabilizing mutations and engineered disulfide bonds, specifically recognized by broadly neutralizing antibodies and resists gp120 conformational change caused by CD4 binding. Injections were administered intramuscularly (IM) and subcutaneously (SC) in a 1 mL volume by needle and syringe. The product was provided at a 500 mcg/mL concentration in 3 mL glass vials filled to 1.2 +/- 0.10 mL. Adjuvant is an aluminum hydroxide suspension (alum) provided in a sterile, pyrogen-free suspension at a concentration of 5 mg/mL in 3 mL glass vials filled to 0.7 +/- 0.10 mL.

Participants:

Healthy adults ages 18 to 50.

Study Plan:

Participants received VRC-HIVRGP096-00-VP at doses of 100 mcg or 500 mcg, both with 500 mcg alum field mixed, administered via IM or SC injections. A dose escalation evaluation occurred to ensure the safety data supported proceeding to the higher dose. Participants were evaluated for safety and immune responses through blood collection at specified timepoints throughout the study.

The study schema is below:

--------------------

Group 1: Participants = 3; Route = IM; Dose (mcg) = 100; Day** 0, Week** 8, Week** 20

Group 2: Participants = 3; Route = SC; Dose (mcg) = 100; Day** 0, Week** 8, Week** 20

Group 3: Participants = 5; Route = IM; Dose (mcg) = 500; Day** 0, Week** 8, Week** 20

Group 4: Participants = 5; Route = SC; Dose (mcg) = 500; Day** 0, Week** 8, Week** 20

Total = 16 Participants

**500 mcg of alum was mixed with Trimer 4571 for all groups

Duration:

Participants were followed for 40 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must have met all of the following criteria:

1. Able and willing to complete the informed consent process.
2. 18-50 years old, inclusive, on day of enrollment.
3. Available for clinic follow-up through the last study visit.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. Willing to donate blood for sample storage to be used for future research.
6. In good general health without clinically significant medical history.
7. Physical examination and laboratory results without clinically significant findings.
8. Body Mass Index (BMI) less than or equal to 40.
9. Assessed as low risk for human immunodeficiency virus (HIV) acquisition by agreeing to discuss HIV infection risks, agreeing to risk reduction counseling, and agreeing to avoid behavior associated with high risk of HIV exposure through the end of study.
10. Screening laboratory values within 56 days prior to enrollment that met the following criteria:

    * Hemoglobin within the institutional normal limits
    * White blood cell (WBC) count between 2,500-12,000/mm^3
    * WBC differential absolute cell counts either within institutional normal range or accompanied by site Principal Investigator (PI) or Associate Investigator (AI) approval, except neutrophils and lymphocytes must specifically be within the range of greater than or equal to 0.75 x the lower limit of normal (LLN) and lees than or equal to 1.25 x the upper limit of normal (ULN) for neutrophil and lymphocyte absolute counts
    * Platelets = 125,000-500,000/m^3
    * Alanine aminotransferase (ALT) less than or equal to 1.25 x ULN based on the institutional normal range
    * Serum creatinine less than or equal to 1.1 x ULN based on the institutional normal range
    * Negative for HIV infection by an FDA approved method of detection

    Woman-specific (if presumed to be of childbearing potential):
11. Agrees to use effective means of birth control from at least 21 days prior to enrollment through the end of the study.
12. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment.

EXCLUSION CRITERIA:

A participant was excluded if one or more of the following conditions apply:

Woman-specific:

1. Breast-feeding or planning to become pregnant through the end of study.

   Participant has received any of the following:
2. An investigational HIV vaccine.
3. Systemic glucocorticoid use equal or greater than prednisone 20mg/day within 4 weeks prior to enrollment, or other medication use likely to impair vaccine response.
4. Blood products within 16 weeks prior to enrollment.
5. Live attenuated vaccines within 4 weeks prior to enrollment.
6. Inactivated vaccines within 2 weeks prior to enrollment.
7. Investigational research agents within 4 weeks prior to enrollment.
8. Current allergen immunotherapy with antigen injections, unless on maintenance schedule.
9. Current anti-tuberculosis (TB) prophylaxis or therapy.

   Participant had any of the following:
10. Serious reactions to vaccines that preclude receipt of study injections as determined by the principal investigator or designee.
11. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
12. Hypertension that is not well controlled.
13. Evidence of significant autoimmune disease or immunodeficiency.
14. Idiopathic urticaria within the past year.
15. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
16. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
17. Asplenia or functional asplenia.
18. Any other chronic or clinically significant condition that in the opinion of the investigator would jeopardize the safety or rights of the study subject including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, psychiatric disorders, heart disease, or cancer.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanders RW, Derking R, Cupo A, Julien JP, Yasmeen A, de Val N, Kim HJ, Blattner C, de la Pena AT, Korzun J, Golabek M, de Los Reyes K, Ketas TJ, van Gils MJ, King CR, Wilson IA, Ward AB, Klasse PJ, Moore JP. A next-generation cleaved, soluble HIV-1 Env trimer, BG505 SOSIP.664 gp140, expresses multiple epitopes for broadly neutralizing but not non-neutralizing antibodies. PLoS Pathog. 2013 Sep;9(9):e1003618. doi: 10.1371/journal.ppat.1003618. Epub 2013 Sep 19. PMID 24068931
- [Background] Kwon YD, Pancera M, Acharya P, Georgiev IS, Crooks ET, Gorman J, Joyce MG, Guttman M, Ma X, Narpala S, Soto C, Terry DS, Yang Y, Zhou T, Ahlsen G, Bailer RT, Chambers M, Chuang GY, Doria-Rose NA, Druz A, Hallen MA, Harned A, Kirys T, Louder MK, O'Dell S, Ofek G, Osawa K, Prabhakaran M, Sastry M, Stewart-Jones GB, Stuckey J, Thomas PV, Tittley T, Williams C, Zhang B, Zhao H, Zhou Z, Donald BR, Lee LK, Zolla-Pazner S, Baxa U, Schon A, Freire E, Shapiro L, Lee KK, Arthos J, Munro JB, Blanchard SC, Mothes W, Binley JM, McDermott AB, Mascola JR, Kwong PD. Crystal structure, conformational fixation and entry-related interactions of mature ligand-free HIV-1 Env. Nat Struct Mol Biol. 2015 Jul;22(7):522-31. doi: 10.1038/nsmb.3051. Epub 2015 Jun 22. PMID 26098315
- [Background] Chuang GY, Geng H, Pancera M, Xu K, Cheng C, Acharya P, Chambers M, Druz A, Tsybovsky Y, Wanninger TG, Yang Y, Doria-Rose NA, Georgiev IS, Gorman J, Joyce MG, O'Dell S, Zhou T, McDermott AB, Mascola JR, Kwong PD. Structure-Based Design of a Soluble Prefusion-Closed HIV-1 Env Trimer with Reduced CD4 Affinity and Improved Immunogenicity. J Virol. 2017 Apr 28;91(10):e02268-16. doi: 10.1128/JVI.02268-16. Print 2017 May 15. PMID 28275193
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. [July 2017]. Available from: https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- [Derived] Houser KV, Gaudinski MR, Happe M, Narpala S, Verardi R, Sarfo EK, Corrigan AR, Wu R, Rothwell RS, Novik L, Hendel CS, Gordon IJ, Berkowitz NM, Cartagena CT, Widge AT, Coates EE, Strom L, Hickman S, Conan-Cibotti M, Vazquez S, Trofymenko O, Plummer S, Stein J, Case CL, Nason M, Biju A, Parchment DK, Changela A, Cheng C, Duan H, Geng H, Teng IT, Zhou T, O'Connell S, Barry C, Carlton K, Gall JG, Flach B, Doria-Rose NA, Graham BS, Koup RA, McDermott AB, Mascola JR, Kwong PD, Ledgerwood JE; VRC 018 Study Team. Safety and immunogenicity of an HIV-1 prefusion-stabilized envelope trimer (Trimer 4571) vaccine in healthy adults: A first-in-human open-label, randomized, dose-escalation, phase 1 clinical trial. EClinicalMedicine. 2022 Jun 1;48:101477. doi: 10.1016/j.eclinm.2022.101477. eCollection 2022 Jun. PMID 35783486
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0031.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland.
Period: Overall Study
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum
Started | 3 | 3 | 5 | 5
Received All Product Administrations | 3 | 3 | 5 | 5
Completed | 3 | 3 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum | Total
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (12.7) | 35.7 (12.5) | 32.4 (8.1) | 32.4 (10.9) | 33.0 (9.7)
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 2 | 1 | 2 | 3 | 8
  31-40 years | 0 | 1 | 2 | 0 | 3
  41-50 years | 1 | 1 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 3 | 10
  Male | 1 | 1 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 2 | 2
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 1 | 3 | 4 | 2 | 10
  Multiracial | 1 | 0 | 1 | 0 | 2
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  Under 18.5 kg/m^2 | 0 | 0 | 1 | 0 | 1
  18.5-24.9 kg/m^2 | 0 | 1 | 2 | 3 | 6
  25.0-29.9 kg/m^2 | 2 | 1 | 2 | 0 | 5
  30.0 kg/m^2 or over | 1 | 1 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms For 7 Days After Each Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after study product administration, at approximately Week 1, Week 9 and Week 21
Population: Population included all enrolled participants who received at least one study product administration and provided safety data (via diary card and/or laboratory results) following study product administration. All participants completed the study product administration schedule per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence Trimer 4571 (100 mcg and 500 mcg): Trimer 4571 dose groups included adults who received either three doses of 100 mcg or three doses of 500 mcg of Trimer 4571 with 500 mcg of alum field mixed administered intramuscularly (IM), or administered subcutaneously (SC) on Day 0, Week 8, and Week 20
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum | Overall Incidence Trimer 4571 (100 mcg and 500 mcg)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Participants
  Pain/Tenderness: None | 1 | 1 | 0 | 0 | 2
  Pain/Tenderness: Mild | 2 | 2 | 5 | 5 | 14
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Swelling: None | 3 | 1 | 4 | 4 | 12
  Swelling: Mild | 0 | 1 | 0 | 0 | 1
  Swelling: Moderate | 0 | 1 | 1 | 1 | 3
  Swelling: Severe | 0 | 0 | 0 | 0 | 0
  Redness: None | 3 | 1 | 4 | 3 | 11
  Redness: Mild | 0 | 0 | 0 | 1 | 1
  Redness: Moderate | 0 | 2 | 1 | 0 | 3
  Redness: Severe | 0 | 0 | 0 | 1 | 1
  Bruising: None | 3 | 3 | 5 | 5 | 16
  Bruising: Mild | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 1 | 1 | 0 | 0 | 2
  Any Local Symptom: Mild | 2 | 0 | 4 | 4 | 10
  Any Local Symptom: Moderate | 0 | 2 | 1 | 0 | 3
  Any Local Symptom: Severe | 0 | 0 | 0 | 1 | 1

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms for 7 Days After Each Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after the study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after study product administration, at approximately Week 1, Week 9 and Week 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum | Overall Incidence Trimer 4571 (100 mcg and 500 mcg)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Participants
  Malaise: None | 3 | 2 | 3 | 3 | 11
  Malaise: Mild | 0 | 0 | 2 | 2 | 4
  Malaise: Moderate | 0 | 1 | 0 | 0 | 1
  Malaise: Severe | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 2 | 3 | 1 | 4 | 10
  Myalgia: Mild | 1 | 0 | 4 | 1 | 6
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0
  Headache: None | 2 | 1 | 4 | 4 | 11
  Headache: Mild | 1 | 2 | 1 | 1 | 5
  Headache: Moderate | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 5 | 5 | 16
  Chills: Mild | 0 | 0 | 0 | 0 | 0
  Chills: Moderate | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0
  Nausea: None | 3 | 2 | 5 | 4 | 14
  Nausea: Mild | 0 | 0 | 0 | 1 | 1
  Nausea: Moderate | 0 | 1 | 0 | 0 | 1
  Nausea: Severe | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 5 | 5 | 16
  Temperature: Mild | 0 | 0 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 2 | 1 | 0 | 2 | 5
  Any Systemic Symptom: Mild | 1 | 1 | 5 | 3 | 10
  Any Systemic Symptom: Moderate | 0 | 1 | 0 | 0 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety
Description: Any abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Labs included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (alanine aminotransferase (ALT) and creatinine). Complete blood count (CBC) with differential, creatine and ALT results were collected at screening, Day 0 prior to the first study product administration (baseline), and Weeks 1-2 after the 1st administration, Week 8 (2nd product administration), and Weeks 9-10 after the 2nd administration, Week 20 (3rd product administration), and Weeks 21-22 after the 3rd administration. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 were used.
Time Frame: Through 40 weeks after the first study product administration
Population: Population included all enrolled participants who had laboratory results available at any study visit post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum | Overall Incidence Trimer 4571 (100 mcg and 500 mcg)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Participants
  ALT | 1 | 0 | 0 | 0 | 1
  Neutrophil count | 0 | 0 | 1 | 0 | 1

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs)
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of each study product administration through the visit scheduled at 28 days (or 4 weeks) after each study product administration. At other time periods greater than the 28-day (or 4-week) post product administration visit, only serious AEs (SAEs reported as a separate outcome and in the AE module), and new chronic medical conditions that required ongoing medical management were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
  If a participant had several AEs and some were evaluated as related and some as unrelated to study product, the participant is counted once as having the related event.
Time Frame: Through 28 days after each study product administration, up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum | Overall Incidence Trimer 4571 (100 mcg and 500 mcg)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Participants
  Related to Study Product | 0 | 2 | 3 | 2 | 7
  Unrelated to Study Product | 1 | 0 | 0 | 1 | 2

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs were recorded from receipt of the study product administration through the last expected study visit at Week 40. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Through 40 weeks after the first study product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum | Overall Incidence Trimer 4571 (100 mcg and 500 mcg)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 16
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Antibody Response to Adjuvanted Trimer 4571 at 2 Weeks After the Final Study Product Administration
Description: Trimer 4571-specific antibody titers were measured by Electrochemiluminescence (ECLIA) using a Meso Scale Discovery (MSD) platform. Serum samples collected at baseline and at 2 weeks after the third product administration were tested in the assay. Since there is no standard/calibration curve available for interpolation of this raw response, area under the curve (AUC) was calculated for each serum sample tested in the 8-fold serial dilutions. The AUC measurement is calculated for each single timepoint sample (baseline or week 22, 2 weeks after the final vaccination). The AUC is calculated with Graphpad Prism™ using the trapezoid rule from the raw sample response (ECL response) over an 8-fold dilution series (Dilution Factor) for each sample. Group geometric mean AUCs and 95% Confidence Intervals are reported.
Time Frame: Baseline through Study Week 22, at 14 days after the final study product administration.
Population: Population included all enrolled participants who received three study product administrations per protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: AUC (ECL response units/Dilution Factor)
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum
Number analyzed (Participants) | 3 | 3 | 5 | 5
AUC (ECL response units/Dilution Factor)
  Antibody Response at Baseline | 81 [40 to 163] | 53 [17 to 169] | 62 [25 to 151] | 50 [26 to 97]
  Antibody Response to Adjuvanted Trimer 4571 at 2 Weeks after the Final Study Product Administration | 674 [50 to 9011] | 924 [175 to 4880] | 2529 [387 to 16515] | 1368 [551 to 3397]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study product administration. Unsolicited AEs were recorded from receipt of each study product administration through the visit scheduled at 28 days (or 4 weeks) after each study product administration. At other time periods greater than the 28-day (or 4-week) post product administration visit, only serious AEs and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: All AEs recorded on the study were reported. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment are reported for participants who received study product and had safety data collected following the product administration. Data represent the number and percentage of participants experiencing the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: Trimer 4571 (100 mcg) IM With Alum | Group 2: Trimer 4571 (100 mcg) SC With Alum | Group 3: Trimer 4571 (500 mcg) IM With Alum | Group 4: Trimer 4571 (500 mcg) SC With Alum
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 5/5 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Trimer 4571 (100 mcg) IM With Alum (N=3) | Group 2: Trimer 4571 (100 mcg) SC With Alum (N=3) | Group 3: Trimer 4571 (500 mcg) IM With Alum (N=5) | Group 4: Trimer 4571 (500 mcg) SC With Alum (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Injection Site Pruritis (General disorders) | 0 | 2 | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Administration site pain (General disorders) | 2 | 2 | 5 | 5
Administration site swelling (General disorders) | 0 | 2 | 1 | 1
Administration site erythema (General disorders) | 0 | 2 | 1 | 2 — Redness
Malaise (General disorders) | 0 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT03783130/Prot_SAP_ICF_000.pdf